CLINICAL TRIAL: NCT02677155
Title: Open Label, Phase II, Study: Sequential Intranodal Immunotherapy (SIIT) Combined With Anti-PD1 (Pembrolizumab) in Patients With Stage III/IV Untreated and Relapsed Follicular Lymphoma
Brief Title: Sequential Intranodal Immunotherapy (SIIT) Combined With Anti-PD1 (Pembrolizumab) in Follicular Lymphoma
Acronym: Lymvac-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Arne Kolstad, MD PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lymvac-2
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Follicular Lymphoma
Keywords: Follicular lymphoma; Intranodal therapy; Autologous dendritic cells; Rituximab; Immunotherapy; Cancer vaccine; Anti-PD1; Pembrolizumab; Radiotherapy
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Radiotherapy; Rituximab; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; pembrolizumab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intranodal immunotherapy and anti-PD1 (Experimental): Induction phase: 3 cycles of sequential intranodal immunotherapy (SIIT), every second week:
  Radiotherapy 8 Gy single dose day 2, Rituximab 5 mg intranodal day 1 and 3, Autologous dendritic cells 1x 10 e8 intranodal day 4 and 5, GM-CSF 50 ug subcutaneously day 4 and 5, Pembrolizumab 200 mg intravenous day 5,
  Consolidation phase:
  Pembrolizumab 200 mg intravenous every third week for 8 cycles
  Interventions: Radiation: Radiotherapy; Biological: Rituximab; Biological: Autologous dendritic cells; Biological: GM-CSF; Biological: Pembrolizumab

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy 8 Gy single dose
Biological: Rituximab — Intranodal injection 5 mg
  Other Names: Mabthera
Biological: Autologous dendritic cells — Intranodal injection of 1 x 10 e8 cells
Biological: GM-CSF — Subcutaneous injection of 50 ug
  Other Names: Sagramostim
Biological: Pembrolizumab — Intravenous infusion of 200 mg
  Other Names: Anti-PD1

SUMMARY:
Follicular lymphoma (FL) is the most common subtype of indolent non-Hodgkin's lymphoma and is often diagnosed in advanced incurable stage. In our previous trail, Lymvac-1, patients were treated with sequential intratumoral injections of low-dose rituximab and autologous dendritic cells, combined with local radiotherapy at the same site. The aim was to overcome tumor tolerance. In this trial, clinical responses correlated strongly with systemic anti-tumor CD8+ T-cell responses detected in blood after therapy. The primary aim of the planned study (Lymvac-2) is to significantly improve rates of immunological and clinical responses by adding iv anti-PD-1 antibody (Pembrolizumab) relative to the cohort of patients previously treated with intranodal immunotherapy without Pembrolizumab (Lymvac-1). The study includes 10 patients with untreated or relapsed FL.

DETAILED DESCRIPTION:
Patients with advanced stage follicular lymphoma, untreated and relapsed are eligible for this study. Staging includes PET/CT, CT and bone marrow specimens. Lymphoma nodes must be available for surgical biopsy, radiation and intranodal treatment. Additionally, there must be evaluable lesions for measuring systemic effects. The patient undergo leukapheresis for collection of monocytes then cultured ex vivo to obtain immature dendritic cells (DC). The treatment targets single lymphoma nodes with radiation (single fraction of 8 Gy), ultrasound-guided injections of autologous DCs , low-dose rituximab (5 mg) and GM-CSF sc. This sequential intranodal immunotherapy (SIIT) is repeated three times, targeting different lymphoma nodes. Anti-PD1 monoclonal antibody (Pembrolizumab) is given iv at each cycle of SIIT and then every third week for a total of 11 cycles. Patients are evaluated for clinical response with PET/CT, CT and bone marrow analysis. CD8 and CD4 T cell responses against autologous tumor cells are measured in blood after treatment by flow cytometry. The primary aims are to induce systemic clinical responses and correlated T cell responses which may prolong time to next standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be >= 18 years of age on day of signing informed consent.
3. Histologically confirmed incurable asymptomatic untreated or relapsed follicular lymphoma grade I-IIIA stage III-IV
4. Lymphoma nodes greater than 1.5 cm at sites suitable for radiation and ultrasound-guided injections
5. Have measurable disease outside irradiated sites.
6. Be willing to provide tissue from an excisional biopsy of a tumor lesion
7. Have a performance status of 0 on the ECOG Performance Scale.
8. Demonstrate adequate organ function as defined below. Absolute neutrophil count (ANC) >=1,500 /mcL, Platelets >=100,000 / mcL, Hemoglobin >=9 g/dL, Serum creatinine >=1.5 X upper limit of normal (ULN) Serum total bilirubin >= 1.5 X ULN. AST (SGOT) and ALT (SGPT) >= 2.5 X ULN OR >= 5 X ULN for subjects with liver metastases, Albumin >=2.5 mg/dL International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) >=1.5 X ULN
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Has progressive lymphoma in need of standard therapy
2. Has transformation to more aggressive disease like diffuse large B cell lymphoma
3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
5. Has a known history of active TB (Bacillus Tuberculosis)
6. Hypersensitivity to rituximab, GM-CSF, pembrolizumab or any of its excipients.
7. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., = Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
8. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., = Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with = Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has known history of, or any evidence of active, non-infectious pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
20. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Evaluated at baseline, 2, 4, 8, 12 and 24 months
  Change in tumor load from baseline until maximal regression

SECONDARY OUTCOMES:
Duration of response | From date of documented response until progression, assessed up to 60 months
  DOR
Progression-free survival | From date of inclusion until date of documented progression or death of any cause, whichever came first, assessed up to 60 months
  PFS
Time to next treatment | From date of inclusion until start of next treatment, assessed up to 60 months
  TNT
Overall survival | From date of inclusion until death of any cause, assessed up to 60 months
  OS
Change in total tumor volume | Compared assessments at inclusion and at time of best response, as assessed up to 60 months, an average of 12 months
  cTTV
Safety: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From inclusion, assessed up to 60 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Anti-tumor T cell responses in blood | Assessed at inclusion and up to 60 months
  T-cell proliferation

CONTACTS AND LOCATIONS:
Overall Officials: Arne Kolstad, MD PhD, Principal Investigator — Dept of Oncology, Oslo University Hospital Radiumhospitalet
Locations (1):
- Oslo University Hospital Radiumhospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Shared when study is published
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After 5 year follow-up
Access Criteria: Collaborating researchers on demand